CLINICAL TRIAL: NCT07196371
Title: Testing the Feasibility of Blood Flow Restriction Training to Enhance the Health Benefits of Exercise in Individuals With Type 2 Diabetes: a Pilot Randomized Controlled Trial
Brief Title: Feasibility of Aerobic Exercise With Blood Flow Restriction Training in People Living With Type 2 Diabetes
Acronym: BOOST-HEALTH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Collaborators: Diabetes Canada (Other); University of Guelph (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Martin Senechal, Full Professor and Acting Assistant Dean of Graduate Studies, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025-069
Record Dates: First submitted 2025-03-13; First posted 2025-09-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Blood flow restriction; aerobic exercise; cardiorespiratory fitness; glycemia; feasability; physical activity; diabetes; continuious glucose monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: single-blind, multi-site, randomized controlled pilot trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training with Blood Flow Restriction (Experimental): Participants will perform aerobic training with blood flow restriction.
  Interventions: Behavioral: Aerobic Training with Blood Flow Restriction
- Standard Aerobic Training (Active Comparator): Participants will perform aerobic training.
  Interventions: Behavioral: Standard Aerobic Training

INTERVENTIONS:
Behavioral: Aerobic Training with Blood Flow Restriction — Participants will undergo a 6-week aerobic training intervention with blood flow restriction applied to the lower limbs.
  Blood flow restriction will be applied using a blood pressure cuff set between 60-80% of limb arterial occlusion pressure.
  Training will consist of treadmill walking at 40-50% of heart rate reserve (HRR) for 32 minutes per session, 3 times per week for a total of 96 minutes per week.
  Arms: Aerobic Training with Blood Flow Restriction
Behavioral: Standard Aerobic Training — Participants will follow the same aerobic training protocol as the AT+BFR group but without blood flow restriction.
  Training will consist of treadmill walking at 40-50% of HRR for 32 minutes per session, 3 times per week for a total of 96 minutes per week.
  Arms: Standard Aerobic Training

SUMMARY:
The goal of this trial is to learn if blood flow restriction training with treadmill walking is possible for individuals living with type 2 diabetes. It will also learn about how the blood flow restriction with treadmill walking could improve health.

The main questions it aims to answer are:

Is 6 weeks of treadmill walking with blood flow restriction reasonable for people with type 2 diabetes to perform? Does treadmill walking with blood flow restriction training help manage type 2 diabetes better than just treadmill walking?

Researchers will compare treadmill walking with blood flow restriction to treadmill walking without blood flow restriction to see if blood flow restriction works to manage type 2 diabetes based on fitness and blood sugar levels.

Participants will:

Perform treadmill walking with or without blood flow restriction for 96 minutes a week for 6 weeks.

Visit the lab before and after the exercise for tests and questionnaires.

DETAILED DESCRIPTION:
Individuals with type 2 diabetes (T2D) display reduced cardiorespiratory fitness, which is a strong predictor of premature mortality and T2D-related complications. Aerobic training (AT) enhances cardiorespiratory fitness and is considered a cornerstone in the management and treatment of T2D. Emerging data suggest that AT combined with blood flow restriction (AT+BFR) training, could potentially enhance cardiorespiratory fitness faster than typical AT in healthy individuals. However, the feasibility of AT+BFR in individuals with T2D and its impact on cardiorespiratory fitness have yet to be determined.

Therefore, the primary objective of this study is to test the feasibility of a 6-week AT+BFR training intervention in individuals with T2D. The secondary objective is to establish preliminary effect sizes for the efficacy of AT+BFR training in individuals with T2D compared to the standard care AT (AT- stdCare).

Methods: This study is a single-blind (investigator & statistical analyst), multi-site, randomized controlled pilot trial of a novel AT+BFR training intervention for individuals living with T2D, which has been informed by patients with lived experience. Participants will be randomized 1:1 using variable permuted block sizes (stratified by sex and site) into 1) AT+BFR or 2) AT-stdCare groups with outcome measures assessed at baseline and 6 weeks.

Population: In 3 sites across Canada, 60 (n=20 per site) individuals living with T2D (5.7% < HbA1c < 9.0%) aged 19-64 years, not meeting the physical activity guidelines (150 mins moderate-vigorous physical activity per week) will be recruited to participate in this 6-week pilot trial.

Intervention: Participants will perform supervised AT+BFR 3 times weekly for 32 minutes per session. A blood pressure cuff will be set between 60-80% of limb arterial occlusion with AT for 96 minutes per week of treadmill walking performed at 40-50% of heart rate reserve (HRR).

Participants in the AT-stdCare will perform 96 minutes per week of treadmill walking at 40-50% of HRR following the same schedule as AT+BFR, training 3 times per week for 32 minutes per session.

Outcomes: The main outcome measures will pertain to the feasibility of a larger trial and include recruitment rates, enrollment and adherence to the intervention, and retention for follow-up testing. The secondary outcomes will be focused on establishing effect sizes to power a larger trial. Effect sizes for the change in cardiorespiratory fitness and continuous glucose monitoring (CGM) outcomes will be determined to help select and power a primary outcome for a more definitive trial of AT+BFR.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes (5.7% < HbA1c < 9.0%)
* Not regularly physically active (150 mins moderate-vigorous physical activity per week)

Exclusion Criteria:

* Musculoskeletal issues preventing exercise training
* Unstable medications over the last 3 months
* Absolute contraindications to BFR (i.e. peripheral vascular disease)
* A self-reported diagnosis of low iron concentrations, anemia, or being treated for these conditions
* A diagnosis of any red blood cell-altering condition (i.e., sickle cell anemia, poikilocytosis)
* Currently living with any cardiovascular disease, which would impact the ability to participate in exercise safely
* Currently prescribed any medication which would impact the ability to use a heart rate monitor to accurately track intensity

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Recruitment | Every 4 weeks up to 2 years
  Recruitment rate will be assessed as the number of individuals who inquire about the trial.
Rate of Enrollment | Every 4 weeks up to 2 years
  Enrollment rate will be assessed as the number of eligible participants who consent to participate in the trial and are randomized to one of the two study arms out of the total number of eligible individuals recruited.
Adherence to the Intervention | From enrollment to the end of intervention at week 6
  Adherence to the intervention will be assessed as the number of sessions that the participant attended out of the total number of sessions.
Rate of Retention for Follow-Up Testing | Every 6 weeks up to 2 years
  Retention rate will be assessed as the number of participants who complete follow-up testing measurements six weeks after randomization.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness (VO2max) | 6 Weeks
  Establishing effect size to power future trials (VO2max)
Glycemia (CGM/HbA1c) | 6 Weeks
  Establishing effect size to power future trials (CGM/HbA1c)
Quality of Life (36-Item Short Form Health Survey (SF-36)) | 6 Weeks
  Establishing effect size to power future trials (SF-36). Scores range from 0-100 for eight domains of health, with higher scores indicating better health-related quality of life and lower scores indicating poorer health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — Cardiometabolic Exercise & Lifestyle Laboratory, Fredericton, New Brunswick
Locations (3):
- Canada (3):
  - Exercise Metabolism and Inflammation Laboratory, Okanagan, British Columbia
  - Cardiometabolic Exercise & Lifestyle Laboratory, Fredericton, New Brunswick
  - Human Performance & Health Research Laboratory, Guelph, Ontario

IPD SHARING:
Plan to Share IPD: Undecided